CLINICAL TRIAL: NCT02653040
Title: Light as an Aid for Recovery in Psychiatric Inpatients: A Pragmatic Randomized Controlled Pilot Trial
Brief Title: Light as an Aid for Recovery in Psychiatric Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QLIGHT
Record Dates: First submitted 2015-12-04; First posted 2016-01-12 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2017-10

CONDITIONS: Mental Illness
Keywords: Lighting; Inpatients; Recovery; Sleep
MeSH Terms: conditions — Mental Disorders | interventions — Lighting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dynamic lighting (Experimental): Indoor lighting with low-lux no-blue wavelengths at night.
  Interventions: Other: Dynamic lighting
- Treatment as usual (No Intervention): Characterized by full white light with little variation through a day cyclus.

INTERVENTIONS:
Other: Dynamic lighting — Intervention is rooms with light settings imitating natural light conditions with white light at day and low-lux no-blue light at night:
  07am-10am: white light, increasing intensity 10am-07pm: white light, full intensity 07pm-11pm: no blue wavelength, low intensity 11pm-07am: no blue wavelength, very low intensity
  Other Names: Illumination, lighting design, lighting environment
  Arms: Dynamic lighting

SUMMARY:
The purpose of this pilot study is to evaluate wether a naturalistic indoor light environment can improve sleep and mood in psychiatric inpatients

DETAILED DESCRIPTION:
Setting: 17 bed inpatient ward at a University Mental Health Hospital

Rooms: The dimensions of all 17 rooms are identical with 4,54m x 3,14m, ceiling height 3,15m, a window, a bed, a table, a chair and a bathroom 1,55m x 1,85m.

Assignment of interventions: After admission patients are invited to participate in the study. If the patients wish to participate they will go through eligibility screen, sign informed consent and fill out questionnaires on sleep, mood and well-being (-t1). The patients (now participants) are randomly allocated (t0) by sealed envelope technique and the envelope is brought to the staff office and opened by a staff member who then from the computer in the office programs the participant's room to either intervention or control.

Randomization: The investigators used random permuted blocks of varying and blinded block size. A third party person created the envelopes and arranged them in blocks.

Blinding: The outcome assessor and data analyst is blinded to allocation. Trial participants and care providers are unblinded. Participants may be replaced to another room for practical, clinical reasons. In this case, the intervention/control conditions will follow the patient.

Data management: All data will be entered in RedCAP and stored in a electronic online secured database at Aarhus University.

Power estimation: Alfa: 0.05. Beta: 0.20. Effect size: change of 4 points in PSQI with a standard deviation estimated to 4. Number of patients in each arm: 17 (x 2 = 34). Number needed to be included accounting for discontinuation: 60 (estimated)

Statistics: The investigators will calculate intention-to-treat. Other statistical analyses will include logistic regression for dichotomous outcome data, analysis of covariance for continuous outcome data, and survival analysis for time-to-event outcome data. Interim-analyses during the data-collection period to stop trial if intervention produces larger than expected benefits or harm or if investigators find evidence of no important difference between experimental and control interventions.

ELIGIBILITY:
Inclusion Criteria:

* Admission

Exclusion Criteria:

* Inability to provide written consent
* Mania

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Sleep quality on the Pittsburgh Sleep Quality Index (PSQI) | Answers from questionnaires are assessed through study completion, an average of 1 month, up to 6 months

SECONDARY OUTCOMES:
Depressive symptoms on the Major depression inventory (MDI) | Answers from questionnaires are assessed through study completion, an average of 1 month, up to 6 months
Well-being on the World Health Organization measure of well-being (WHO-5) | Answers from questionnaires are assessed through study completion, an average of 1 month, up to 6 months
Qualitative assessment using a custom made questionnaire | Answers from questionnaires are assessed through study completion, an average of 1 month, up to 6 months
  Number of patients with side-effects.
Sleep diary | Answers from questionnaires are assessed through study completion, an average of 1 month, up to 6 months

OTHER OUTCOMES:
Time to discharge | Assessed through study completion, an average of 1 month, up to 6 months
  Number of days between admission and discharge
Involuntary restraints | Assessed through study completion, an average of 1 month, up to 6 months
  Number of participants who experienced involuntary physical and/or medical restraints.
Use of medication from logged activity in the electronic medical record | Assessed through study completion, an average of 1 month, up to 6 months
  Use of medication during admission including drug og dosages administered to the participants in mg/day.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Okkels, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Affective Disorders, Aarhus University Hospital, Risskov, Risskov, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bedrosian TA, Nelson RJ. Influence of the modern light environment on mood. Mol Psychiatry. 2013 Jul;18(7):751-7. doi: 10.1038/mp.2013.70. Epub 2013 May 28. PMID 23711982
- [Background] LeGates TA, Fernandez DC, Hattar S. Light as a central modulator of circadian rhythms, sleep and affect. Nat Rev Neurosci. 2014 Jul;15(7):443-54. doi: 10.1038/nrn3743. Epub 2014 Jun 11. PMID 24917305